CLINICAL TRIAL: NCT05208866
Title: PA-ADPKD-304: A Phase 3, Open-label, Roll-over Study to Assess Long-term Safety of Lixivaptan in Participants With Autosomal Dominant Polycystic Kidney Disease Who Completed Study PA-ADPKD-303: The ALERT Study
Brief Title: Roll-over Study to Assess Safety of Lixivaptan in Participants With ADPKD Who Completed Study PA-ADPKD-303
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: The decision is based on a thorough reassessment of the commercial potential of lixivaptan as a potential best-in-class therapy for patients with ADPKD.
Sponsor: Palladio Biosciences (Industry)
Collaborators: Centessa Pharmaceuticals plc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PA-ADPKD-304
Record Dates: First submitted 2022-01-07; First posted 2022-01-26 (Actual); Results first posted 2023-04-10 (Actual); Last update posted 2023-05-12 (Actual); Status verified 2023-04

CONDITIONS: Polycystic Kidney Disease, Adult
MeSH Terms: conditions — Polycystic Kidney, Autosomal Dominant | interventions — lixivaptan

STUDY DESIGN:
Intervention Model Description: Single group, open-label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Lixivaptan (Experimental): Lixivaptan capsules 100-200mg twice daily
  Interventions: Drug: Lixivaptan

INTERVENTIONS:
Drug: Lixivaptan — Oral vasopressin V2 receptor antagonist

SUMMARY:
This is a Phase 3, open-label, roll-over study to demonstrate the continued hepatic and non-hepatic safety and renal efficacy of lixivaptan in participants with ADPKD who previously experienced abnormal liver chemistry test results while treated with tolvaptan, were permanently discontinued from the drug for that reason, and subsequently completed study PA-ADPKD-303, the open-label lead-in study with lixivaptan.

DETAILED DESCRIPTION:
This is a Phase 3, open-label, roll-over study to demonstrate the continued hepatic and non-hepatic safety and renal efficacy of lixivaptan in participants with ADPKD who previously experienced abnormal liver chemistry test results while treated with tolvaptan that resulted in permanent discontinuation of tolvaptan for that reason, and subsequently completed study PA-ADPKD-303, the open-label lead-in study with lixivaptan.

Assessments completed during the final 4 visits of PA-ADPKD-303, the lead-in study, will serve as the screening and baseline assessments for this roll-over study. Evaluation of eligibility will be completed at Visit 1 of this study, following signing of informed consent. Participants satisfying all study entry criteria at Visit 1 will be considered enrolled following completion of all Visit 1 study procedures and will be dispensed lixivaptan treatment to start the Lixivaptan Re-titration Period (1 to 2 weeks). During the Lixivaptan Re-titration Period, participants will have their dose of lixivaptan re-established based on the dose they were receiving at the completion of the lead-in study. Participants will continue on lixivaptan treatment for up to 104 weeks during the Maintenance Treatment Period and will be assessed at a study visit every 12 weeks. In between the quarterly study visits, participants will be required to have blood drawn for liver chemistry determinations every 4 weeks. At the end of 104 weeks, lixivaptan treatment will be stopped, and participants will enter a 4-week Follow-up Period during which final assessments of safety and efficacy will be obtained over 3 visits during a 28-day period.

ELIGIBILITY:
Inclusion Criteria:

* Male or female participants with ADPKD who completed study PA-ADPKD-303
* Continued control of hypertension without the use of a diuretic
* Continued adherence to prohibitions on concomitant medications stated in the study PA-ADPKD-303 protocol
* Willing to practice acceptable methods of birth control (both males who have partners of child-bearing potential and females of childbearing potential).
* Able to provide informed consent.

Exclusion Criteria:

* Any contraindication to continued treatment with lixivaptan
* Clinically significant incontinence, overactive bladder, or urinary retention (e.g., benign prostatic hyperplasia)
* New York Heart Association Functional Class 3 or 4 heart failure or other significant cardiac or electrocardiogram (ECG) findings that could pose a safety risk to the participant
* Hypovolemia on physical examination at Screening
* The following laboratory results based on serum drawn at Visit 24 of PA-ADPKD-303:

  * Serum alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values >1.5 × ULN
  * Total bilirubin values >1.5 × ULN
* eGFR <20 mL/min/1.73 m^2 based on laboratory results from Visit 26 of PA-ADPKD-303
* A finding at Screening that precludes safe participation in the study or participants who are likely to be non-compliant with study procedures in the opinion of the Investigator or medical monitor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2022-02-10 (Actual); Primary Completion 2022-06-29 (Actual); Study Completion 2022-07-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nelson Kopyt, DO, Principal Investigator — Northeast Clinical Research Center, LLC
Locations (1):
- Northeast Clinical Research Center, LLC, Bethlehem, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fontana RJ, Watkins PB, Bonkovsky HL, Chalasani N, Davern T, Serrano J, Rochon J; DILIN Study Group. Drug-Induced Liver Injury Network (DILIN) prospective study: rationale, design and conduct. Drug Saf. 2009;32(1):55-68. doi: 10.2165/00002018-200932010-00005. PMID 19132805

RESULTS

PARTICIPANT FLOW:
Groups:
- All Enrolled Participants: All participants who were enrolled in this study were included in this group.
Period: Lixivaptan Re-titration Period
Arm/Group | All Enrolled Participants
Started | 1
Completed | 1
Not Completed | 0
Period: Maintenance Treatment Period
Arm/Group | All Enrolled Participants
Started | 1
Completed | 0
Not Completed | 1
Not completed — Sponsor Termination of Study | 1
Period: Follow-up Period
Arm/Group | All Enrolled Participants
Started | 1 (All participants who were treated with lixivaptan completed the Follow-up Period, including those who did not complete the Maintenance Period.)
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Since only one participant completed the study, due to confidentiality issues, no data will be reported.
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 0
Age, Continuous [unit: Years]
Sex: Female, Male
Ethnicity (NIH/OMB)
Race (NIH/OMB)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Who Develop Serum ALT Levels >3 × ULN During the Lixivaptan Re-titration or Maintenance Treatment Periods Assessed to be Related to Lixivaptan and Resulted in Discontinuation of Lixivaptan Treatment
Description: Number of participants who develop serum alanine aminotransferase (ALT) levels >3 × the upper limit of normal (ULN) which are assessed by the independent Hepatic Events Review Committee (HERC) to be at least probably related to lixivaptan and resulted in discontinuation of lixivaptan treatment. The independent HERC, after reviewing demographic, medical and medication history, safety data and other relevant data of participants who develop liver abnormalities, will determine the probable causality for liver chemistry test abnormalities of concern and the relatedness to lixivaptan using the Drug-Induced Liver Injury Network probability criteria (Fontana et al., 2009). The normal range of ALT was defined as 0-55 U/L.
Time Frame: 120 days (from Screening to the end of the Maintenance Treatment Period)
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1
Participants | 0

2. Secondary Outcome: Number of Participants Who Develop Serum ALT Levels >5 x ULN During the Lixivaptan Re-titration or Maintenance Treatment Periods Assessed to be Related to Lixivaptan and Resulted in Discontinuation of Lixivaptan Treatment
Description: Number of participants who develop serum ALT levels >5 × ULN which are assessed by the independent HERC to be at least probably related to lixivaptan and resulted in discontinuation of lixivaptan treatment. The independent HERC, after reviewing demographic, medical and medication history, safety data and other relevant data of participants who develop liver abnormalities, will determine the probable causality for liver chemistry test abnormalities of concern and the relatedness to lixivaptan using the Drug-Induced Liver Injury Network probability criteria (Fontana et al., 2009). The normal range of ALT was defined as 0-55 U/L.
Time Frame: 120 days (from Screening to the end of the Maintenance Treatment Period)
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1
Participants | 0

3. Secondary Outcome: Number of Participants Who Develop Serum ALT Values >3 × ULN During the Lixivaptan Re-titration or Maintenance Treatment Periods Assessed to be Related to Lixivaptan and Resulted in Dose Reduction of Lixivaptan Treatment
Description: Number of participants who develop serum ALT levels >3 × ULN that were assessed by the independent HERC to be at least probably related to lixivaptan and resulted in dose reduction of lixivaptan treatment. The independent HERC, after reviewing demographic, medical and medication history, safety data and other relevant data of participants who develop liver abnormalities, will determine the probable causality for liver chemistry test abnormalities of concern and the relatedness to lixivaptan using the Drug-Induced Liver Injury Network probability criteria (Fontana et al., 2009). The normal range of ALT was defined as 0-55 U/L.
Time Frame: 120 days (from Screening to the end of the Maintenance Treatment Period)
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1
Participants | 0

4. Secondary Outcome: Number of Participants With Treatment-emergent Adverse Events (TEAEs)
Description: Number of participants with TEAEs during the Lixivaptan Re-titration Period, the Maintenance Treatment Period, or the Follow-up Period.
Time Frame: 140 days (from Screening to the end of the Follow-up Period)
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1
Participants
  Lixivaptan Re-titration and Maintenance Treatment Periods | 1
  Follow-up Period | 0

5. Secondary Outcome: Number of Participants With Potentially Clinically Important Clinical Laboratory Findings
Description: Number of participants with clinical laboratory findings (non-hepatic clinical chemistry, hematology, and urinalysis) recorded during the Lixivaptan Re-titration Period, the Maintenance Treatment Period, or the Follow-up Period, and considered to be potentially clinically important.
Time Frame: 140 days (from Screening to the end of the Follow-up Period)
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1
Participants
  Lixivaptan Re-titration and Maintenance Treatment Periods | 0
  Follow-up Period | 0

6. Secondary Outcome: Number of Participants With Potentially Clinically Important Vital Signs Findings
Description: Number of participants with vital signs findings (heart rate, diastolic and systolic blood pressure, and weight) recorded during the Lixivaptan Re-titration Period, the Maintenance Treatment Period, or the Follow-up Period, and considered to be potentially clinically important.
Time Frame: 140 days (from Screening to the end of the Follow-up Period)
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1
Participants
  Lixivaptan Re-titration and Maintenance Treatment Periods | 0
  Follow-up Period | 0

7. Secondary Outcome: Number of Participants With Potentially Clinically Important 12-lead Electrocardiogram (ECG) Findings
Description: Number of participants with ECG findings recorded during the Lixivaptan Re-titration Period, the Maintenance Treatment Period, or the Follow-up Period, and considered to be potentially clinically important (defined as a QT interval corrected for heart rate according to Fridericia's formula [QTcF] ≥ 450 msec).
Time Frame: 140 days (from Screening to the end of the Follow-up Period)
Measure: Count of Participants; unit: Participants
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1
Participants
  Lixivaptan Re-titration and Maintenance Treatment Periods | 0
  Follow-up Period | 0

8. Secondary Outcome: Annualized Change in Estimated Glomerular Filtration Rate (eGFR) From Baseline to Final Assessment
Description: Baseline eGFR is defined as the mean of the 3 eGFR assessments obtained at Visits 25, 26 and 27 of study PA-ADPKD-303 (if any values are missing, the remaining values will be used to determine the baseline eGFR). The endpoint eGFR is defined as the mean of 3 eGFR assessments obtained during the Follow-up Period (if any values are missing, the remaining values will be used to determine the endpoint eGFR). The change in eGFR from Baseline to Final Assessment will be provided.
Time Frame: 140 days (from Screening to the end of the Follow-up Period)
Population: The annualized change in eGRF is provided for the only participant enrolled at the time of early termination of the study.
Measure: Mean (Standard Deviation); unit: mL/min/1.73m^2
Arm/Group | All Enrolled Participants
Number analyzed (Participants) | 1
mL/min/1.73m^2 | 14.6 (0.0)

ADVERSE EVENTS:
Time Frame: Adverse events were recorded from when participants had taken their first dose of lixivaptan in the Re-titration Period until the end of the study (maximum duration: 140 days)
Groups:
- Titration and Maintenance Periods: All participants who completed the Lixivaptan Re-titration Period and entered the Maintenance Period
- Follow-up Period: All participants who entered the Follow-up Period, regardless of whether they had completed the Maintenance Period
Arm/Group | Titration and Maintenance Periods | Follow-up Period
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/1
Other Adverse Events (participants affected / at risk) | 1/1 | 0/1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Titration and Maintenance Periods (N=1) | Follow-up Period (N=1)
Dermatitis contact (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0)
Arthropod bite (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
Efficacy and safety results are limited by the early termination of the trial and the small number of subjects. Early termination was due to a sponsor decision for reasons unrelated to safety.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of more than 60 days

DOCUMENTS (2):
  • Study Protocol (2022-05-20): https://cdn.clinicaltrials.gov/large-docs/66/NCT05208866/Prot_000.pdf
  • Statistical Analysis Plan (2022-09-24): https://cdn.clinicaltrials.gov/large-docs/66/NCT05208866/SAP_001.pdf